CLINICAL TRIAL: NCT01814761
Title: A Study of Bimatoprost 0.01% in the Clinical Setting
Acronym: APPEAL-Taiwan
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-AP-EYE-AGN-001
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Results first posted 2015-10-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-09

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pts with POAG or OH (Previously Treatment Naive): Previously treatment naïve patients with Primary Open-Angle Glaucoma (POAG) or Ocular Hypertension (OH) who require treatment with bimatoprost 0.01% (Lumigan® 0.01%).
  Interventions: Drug: Bimatoprost 0.01%
- Pts with POAG or OH (Switched Monotherapy): Patients previously on another monotherapy treatment with Primary Open-Angle Glaucoma (POAG) or Ocular Hypertension (OH) who require treatment with bimatoprost 0.01% (Lumigan® 0.01%).
  Interventions: Drug: Bimatoprost 0.01%

INTERVENTIONS:
Drug: Bimatoprost 0.01% — One drop of bimatoprost 0.01% (Lumigan® 0.01%) in the affected eye(s) every evening for 12 weeks.
  Other Names: Lumigan® 0.01%

SUMMARY:
This is a study of bimatoprost 0.01% (LUMIGAN® 0.01%) in subjects with primary open-angle glaucoma (POAG) or ocular hypertension (OH) who require further treatment for elevated intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma or ocular hypertension
* Determined by the treating physician to require treatment with bimatoprost 0.01%.

Exclusion Criteria:

* Previous use of Lumigan® 0.01%

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with primary open-angle glaucoma or ocular hypertension
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2013-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Taichung, Taiwan

REFERENCES:
- [Derived] Chen YY, Wang TH, Liu C, Wu KY, Chiu SL, Simonyi S, Lu DW. Tolerability and efficacy of bimatoprost 0.01 % in patients with open-angle glaucoma or ocular hypertension evaluated in the Taiwanese clinical setting: the Asia Pacific Patterns from Early Access of Lumigan 0.01 % (APPEAL Taiwan) study. BMC Ophthalmol. 2016 Sep 15;16(1):162. doi: 10.1186/s12886-016-0338-6. PMID 27633513

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pts With POAG or OH (Previously Treatment Naive) | Pts With POAG or OH (Switched Monotherapy)
Started | 42 | 270
Completed | 34 | 240
Not Completed | 8 | 30
Not completed — Other Reasons | 1 | 10
Not completed — Ocular Adverse Event | 6 | 15
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pts With POAG or OH (Previously Treatment Naive) | Pts With POAG or OH (Switched Monotherapy) | Total
Number analyzed (Participants) | 42 | 270 | 312
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (13.65) | 53.4 (14.45) | 53.3 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 114 | 134
  Male | 22 | 156 | 178

OUTCOME MEASURES:

1. Secondary Outcome: Change From Baseline in Intraocular Pressure (IOP) in the Study Eye
Description: IOP is a measure of the fluid pressure inside the eye. A negative number change from baseline indicates a reduction in IOP (improvement) and a positive number change from baseline indicates an increase in IOP (worsening).
Time Frame: Baseline, Week 12
Population: Intent-to-Treat: Enrolled patients who received at least one dose of study medication and who were not currently treated with Bimatoprost 0.01% at the time of enrollment
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Pts With POAG or OH (Previously Treatment Naive) | Pts With POAG or OH (Switched Monotherapy)
Number analyzed (Participants) | 42 | 270
Millimeters of Mercury (mmHg)
  Baseline | 18.0 (3.82) | 17.8 (3.89)
  Week 12 (N=34, 240) | -3.6 (3.55) | -2.6 (3.22)

2. Secondary Outcome: Percentage of Patients Who Discontinue Due to an Adverse Event
Description: An adverse event is any untoward medical occurrence associated with the use of a drug, whether or not considered drug related.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Number; unit: Percentage of Patients
Arm/Group | Pts With POAG or OH (Previously Treatment Naive) | Pts With POAG or OH (Switched Monotherapy)
Number analyzed (Participants) | 42 | 270
Percentage of Patients | 14.3 | 5.6

3. Primary Outcome: Severity of Ocular Hyperemia in the Study Eye on a 5-Point Scale
Description: Hyperemia is the engorgement of the blood vessels (redness) of the eye. Hyperemia is graded in the study eye on a 5-point scale where 0=None (Normal), 0.5=Trace (Trace reddish pink with no more than slight perilimbal injection), 1=Mild (Mild flush reddish color), 2=Moderate (Bright red color), and 3=Severe (Deep, bright, diffuse redness). The numbers of patients in each severity grade are presented.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Number; unit: Patients
Arm/Group | Pts With POAG or OH (Previously Treatment Naive) | Pts With POAG or OH (Switched Monotherapy)
Number analyzed (Participants) | 42 | 270
Patients
  None | 7 | 36
  Trace | 10 | 50
  Mild | 12 | 84
  Moderate | 5 | 59
  Severe | 0 | 11
  Missing | 8 | 30

4. Secondary Outcome: Overall Percent Change From Baseline in IOP
Description: IOP is a measure of the fluid pressure inside the eye. A negative number change response indicates a reduction in IOP (improvement) and a positive number change response indicates an increase in IOP (worsening).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Pts With POAG or OH (Previously Treatment Naive) | Pts With POAG or OH (Switched Monotherapy)
Number analyzed (Participants) | 34 | 240
Percentage Change | -19.25 [-24.8 to -13.7] | -13.26 [-15.4 to -11.2]

ADVERSE EVENTS:
Description: The Safety Population is used to assess serious adverse events (SAEs) and adverse events (AEs) and included all enrolled patients who received at least one dose of study medication and who were not currently treated with Bimatoprost 0.01% at the time of enrollment (same as the intent-to-treat population)
Arm/Group | Pts With POAG or OH (Previously Treatment Naive) | Pts With POAG or OH (Switched Monotherapy)
Serious Adverse Events (participants affected / at risk) | 1/42 | 2/270
Other Adverse Events (participants affected / at risk) | 10/42 | 16/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pts With POAG or OH (Previously Treatment Naive) (N=42) | Pts With POAG or OH (Switched Monotherapy) (N=270)
Urinary Tract Infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Intracranial Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pts With POAG or OH (Previously Treatment Naive) (N=42) | Pts With POAG or OH (Switched Monotherapy) (N=270)
Ocular Hyperaemia (Eye disorders) | 7 | 14
Dry Eye (Eye disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.